CLINICAL TRIAL: NCT01139268
Title: Examination of Gene Expression, Time-lapse and Near-infrared Spectroscopy (NIR) to Identify Differences in Embryo Viability
Brief Title: Identification of Viable Human Embryos Using Three Different Methods
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: M-20090241
Record Dates: First submitted 2010-06-07; First posted 2010-06-08 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Infertility
Keywords: embryo viability
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — biopsies from human embryos
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Infertility affects an increasing number of couples. For many, the choice of treatment is in vitro fertilization (IVF) . Currently, there are no markers fully predictive of developmental competence of IVF embryos. Present embryo selection is based on morphology assessment, which produces implantation rates in the range of 20%-30 %. The overall purpose of the present study is to investigate methods for selection of the best embryo. We aim to examine the relationship between pregnancy outcome and the transcriptional profile of selected genes, cleavage kinetics (time-lapse), and metabolic profile. We hypothesise that the quality of the embryo is reflected by the transcription of selected genes, the cleavage kinetics, and the metabolic profile. If so, these parameters can predict the success or failure of a pregnancy. Furthermore, the interrelationship - if any - between these parameters will be evaluated.

A secondary aim is to evaluate the effect of blastomere biopsy using time-lapse and metabolic analysis

DETAILED DESCRIPTION:
Introduction:

Infertility affects an increasing number of couples. For many, the choice of treatment is In Vitro Fertilization (IVF). Currently, there are no markers fully predictive of developmental competence of human IVF embryos. Present embryo selection is based on morphology assessment, which produces implantation rates in the range of 20-30 %. To maximize the probability of obtaining a pregnancy, multiple embryos are often transferred simultaneously at the risk of multiple gestations. The high multiple pregnancy rates associated with IVF increases the risk of neonatal complications and maternal pregnancy-related health problems. Single Embryo Transfer (SET) is an effective way of minimizing the risk of multiple gestations, but an accurate method of selecting the most viable embryo will optimise the use of SET. Today, the quality of an embryo is assessed using microscopic evaluation of morphological parameters, but the method has limited predictive value. Therefore, several areas are investigated in search of additional markers of viability in order to reduce multiple gestation rates and improve implantation rates, but all have yet to prove their value in a clinical setting.

Gene expression profiling is a novel strategy with potential to identify the most viable embryo. Several publications suggest that differences in gene expression patterns are related to embryo potential and quality. A bovine study identified specific genes related to viability using microarray technology, proposing their use as markers of viability. A similar study has been performed on human embryos, identifying 7000 transcripts associated to successful IVF treatment.

Time-lapse analysis is another way of assessing embryo potential. Studying cleavage kinetics, where milestones of early development, such as fertilization, cleavage, synchrony and duration of cleavage, are correlated to differences in time intervals, might very well be a useful marker of embryo viability. Recently, an EmbryoScope (Unisense Fertitech, http://www.unisense.com/Default.aspx?ID=170) has been developed that allows series of photos taking during incubation (Time-lapse). The pictures are taken every 30 minutes within a controlled incubator housed with camera and microscope

Embryo metabolism is considered a critical determinant of viability, and it is likely that viable embryos possess a unique metabolic profile, expressed by composition of metabolites in the culture medium. Metabolomics studies the inventory of metabolites representing the functional genotype. Near-Infrared (NIR) spectroscopy is an analytic technique based on spectroscopy in the near infrared region suitable for rapid analysis of the metabolome. Recent publications suggest that the metabolic profile can be used to identify high potential embryos using NIR .

Aim and hypothesis. The purpose of the present study is to examine pregnancy outcome/potential to implant and its relationship to 1) transcriptional profile of selected genes,, 2) cleavage kinetics, and 3) metabolic profile. In particular we hypothesize that the transcription of selected genes, the cleavage kinetics and the metabolic profile from embryos with high developmental competence and implantation potential will differ from embryos of lower quality and therefore that these parameters will be predictive of pregnancy success. Furthermore, the interrelationship - if any - between these parameters will be evaluated.

A secondary aim is to evaluate the effect of blastomere biopsy using time-lapse and metabolic analysis

Perspective: Should the analysis of selected genes, Time-Lapse or metabolic profiles prove predictive of viability, the methods could be used supplementary when assessing embryo viability, refining the existing criteria. Apart from generating new knowledge concerning the biology of the preimplantation embryo, the study aims to improve existing IVF techniques.

1. Bioinformatical and comparative examination of homology and transcription in bovine and human genes; identification of human candidate genes Purpose: To identify human analogues to the 52 bovine candidate genes by comparing nucleotide sequences and gene transcription between humans and cattle, using databases and bioinformational tools. Based on the results and existing publications and knowledge concerning gene expression and embryogenesis in humans and cattle 12 genes will be selected for further analysis. After designing primers for RT-PCR, ultra sensitive, quantitative (q)-rt-PCR analyses are developed. Before testing humane embryos, the analyses will be performed on human cell-lines.

   Materials and methods: In brief, cells are lysed and mRNA isolated, using an mRNA extraction kit. cDNA is generated using reverse transcriptase PCR with sequence specific primers. Quantitative analyses of embryo cDNA are performed with Real Time PCR on Roche Light-cycler using fluorescence DNA labelling. Results are reported as relative expressions to an endogenous control.
2. Quantification and variation of putative pregnancy-related genes in biopsies from human blastocysts Purpose: Quantification of max. 12 selected genes on biopsies from humane IVF blastocysts using RT-PCR and Real-Time PCR. The results will be used to select 5 genes for further analysis. The main purpose is to characterize and describe variations in transcription of the selected genes in human preimplantation embryos.

Materials and methods Couples undergoing IVF treatment in order to permit preimplantation genetic diagnosis (PGD) of the embryo will be requested permission to include embryos with diagnosed gene or chromosomal disorders in the project, embryos which under normal circumstances are discarded. The diagnosis healthy/diseased is made by PCR og FISH analysis of a blastomere biopsied on day 3 (8-cell stage). The embryos are routinely cultured in the EmbryoScope until day 5 after oocyte retrieval.

Embryo biopsy Embryos included in the project are cultured until day 5 after oocyte retrieval. On day 3 the embryos are biopsied using a laser. The biopsies are marked and frozen for later analysis.

Gene expression analysis The gene expression in cells from the biopsies are analysed using RT-PCR and real-time PCR as described (project 1) with the purpose of quantifying 2-5 genes from each individual cell, quantifying at maximum 12 genes. Each gene is analysed in biopsies from 10 different embryos, to characterize inter-individual differences. From each blastocyst are taken at least two biopsies, which are subjected to identical RT-PCR and rt-PCR analyses to evaluate potential intra-individual differences and to validate the method.

Time-lapse analysis: Embryos are cultured in the EmbryScope, images are recorded every 20 min.

3A, B and C: Implantation in relation to transcription of selected genes, Time-Lapse parameters, and metabolic profile Purpose: To correlate result of the IVF treatment (+/- clinical pregnancy) to A: the expression of 5 selected genes B: cleavage kinetics using Time-Lapse analysis C: metabolic profile using Near-Infrared (NIR) Spectroscopy

Culturing of embryos In Denmark, IVF embryos are currently normally transferred 2-3 days after oocyte retrieval.. Improvements of media techniques used for culturing have led to a trend towards blastocyst transfer in many clinics. During the first week of preimplantation development, gene transcription switch from maternal to embryonic control, and the energy metabolism changes. Furthermore, the proportion of euploid embryos is higher when comparing blastocysts with cleavage stage embryos. On the other hand, some embryos arrest their development, leaving fewer embryos available for transfer. The latest Cochrane (2007) analysis concludes that there is growing evidence in favour of blastocyst transfer for SET, in particular when treating women with many retrieved oocytes. Genetic material from the embryo can be obtained by performing biopsies on either the cleavage-stage embryo (8 cells), where one or two blastomeres are removed, or from the blastocyst (about 100 cells), taking 2-10 cells from the trophectoderm (TE). Advantages of TE biopsy include obtaining more genomic material (DNA/RNA), which improves the diagnostic reliability. The embryo is exposed to less stressful conditions, since a relatively smaller proportion of cells is removed, plus the biopsy is performed from extra-embryonic tissue, that is, cells forming the placenta. Blastocyst biopsy does not appear to impair developmental competence and implantation (13,17-19). In conclusion, performing TE biopsy on blastocysts seems to be less invasive and stressful while yielding more information, thus making it our choice of method.

Biopsy On day 3 after oocyte retrieval, a small hole in zona pellucida is made with a laser, allowing the TE to herniate through the hole during the next 2 days incubation. Early on day 5 embryos are assessed for blastocyst development according to the criteria listed below, and one embryo is chosen for transfer. TE biopsy is performed on this embryo by aspirating the herniating TE, approximately 2-20 cells, into an embryo biopsy pipette and cutting it off with laser. The cells are immediately frozen for later analysis. The spent embryo medias are collected individually and frozen at - 80 C for later NIR analysis. Models of spectral regions are used to calculate an individual viability index for each embryo. Urine hCG test and ultrasound at gestational ages 8 and 12 are used to determine pregnancy outcome.

Blastocyst score: Embryos are evaluated on day 5 using criteria described by Gardner et al, where blastocyst are scored according to size. Briefly, the blastocysts were graded according to size: [1] early blastocyst, the blastocoel is less than half the volume of the embryo; [2] blastocyst, the blastocoel is greater than or equal to half of the volume of the embryo; [3] full blastocyst, the blastocoel completely fills the embryo; [4] expanded blastocyst, the blastocoel volume is larger than that of the early embryo and the zona is thinning; [5] hatching blastocyst, the trophectoderm has started to herniate through the zona; and [6] hatched blastocyst, the blastocyst has completely escaped from the zona. For blastocysts graded as 3 to 6 (i.e., full blastocysts and onward) the development of the inner cell mass (ICM) and trophectoderm can be assessed. The ICM grading is as follows: A. tightly packed, many cells; B. loosely grouped, several cells; C. very few cells. The trophectoderm grading is as follows: A. many cells forming a tightly knit epithelium; B. few cells; C. very few cells forming a loose epithelium.

ELIGIBILITY:
Inclusion Criteria:

* age < 38 years
* > 8 retrieved oocytes in present cycle or > 6 fertilized.

Exclusion Criteria:

* endometriosis

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women undergoing ART treament with single embryo transfer at the Fertility clinic, Aarhus University hospital Skejby, due to infertility,
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2010-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
implantation/clinical pregnancy confirmed with pregnancy test and ultrasound | 8 weeks after embryo transfer
  measurement of urine-hCG and vaginal ultrasound scan to evaluate pregnant/not pregnant

SECONDARY OUTCOMES:
gene expression quantified with Q-PCR | within 6 months after biopsy and embryo transfer
  RT-Q-PCR analysis of selected genes
Metabolic profile using NIR analysis | within 6 months after collection
  Near Infrared Spectroscopy (NIR) of the spent culture media. The spectral profile is used to calculate a viability index
cleavage kinetics | before embryo transfer, during culturing
  imaging of the developing embryos during culturing. Data analysis concerning morphological parametres within 6 months after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Ingerslev, MD, DMsc, Study Director — Fertility Clinic, Aarhus University Hospital, Skejby; kirstine Kirkegaard, MD, Principal Investigator — Fertility Clinic, Aarhus University Hospital, Skejby; Johnny Hindkjær, DM.Sc., Principal Investigator — Fertility Clinic, Aarhus University Hospital, Skejby; Birte Degn, DmSc. PhD, Principal Investigator — Fertility Clinic, Aarhus University Hospital, Skejby; Karin Lykke-Hartmann, DmSc, PhD, Principal Investigator — Aarhus University, Department of Medical Biochemistry; Steen Koelvraa, MD, DMSc, Principal Investigator — Department of Clinical Genetics, Vejle Hospital
Locations (2):
- Denmark (2):
  - The Fertility Clinic, Aarhus University Hospital, Skejby, Aarhus
  - Fertility Clinic, Aarhus University Hospital Skejby, Aarhus N

REFERENCES:
- [Derived] Kirkegaard K, Svane AS, Nielsen JS, Hindkjaer JJ, Nielsen NC, Ingerslev HJ. Nuclear magnetic resonance metabolomic profiling of Day 3 and 5 embryo culture medium does not predict pregnancy outcome in good prognosis patients: a prospective cohort study on single transferred embryos. Hum Reprod. 2014 Nov;29(11):2413-20. doi: 10.1093/humrep/deu236. Epub 2014 Sep 24. PMID 25256566
- [Derived] Sundvall L, Ingerslev HJ, Breth Knudsen U, Kirkegaard K. Inter- and intra-observer variability of time-lapse annotations. Hum Reprod. 2013 Dec;28(12):3215-21. doi: 10.1093/humrep/det366. Epub 2013 Sep 26. PMID 24070998
- [Derived] Kirkegaard K, Hindkjaer JJ, Ingerslev HJ. Hatching of in vitro fertilized human embryos is influenced by fertilization method. Fertil Steril. 2013 Nov;100(5):1277-82. doi: 10.1016/j.fertnstert.2013.07.005. Epub 2013 Jul 30. PMID 23909991
- [Derived] Kirkegaard K, Kesmodel US, Hindkjaer JJ, Ingerslev HJ. Time-lapse parameters as predictors of blastocyst development and pregnancy outcome in embryos from good prognosis patients: a prospective cohort study. Hum Reprod. 2013 Oct;28(10):2643-51. doi: 10.1093/humrep/det300. Epub 2013 Jul 30. PMID 23900207
- [Derived] Kirkegaard K, Hindkjaer JJ, Ingerslev HJ. Effect of oxygen concentration on human embryo development evaluated by time-lapse monitoring. Fertil Steril. 2013 Mar 1;99(3):738-744.e4. doi: 10.1016/j.fertnstert.2012.11.028. Epub 2012 Dec 11. PMID 23245683